CLINICAL TRIAL: NCT00924404
Title: Randomized Controlled Trial of Xylitol Versus Saline Rinse For Chronic Sinusitis
Brief Title: Xylitol Versus Saline in Chronic Sinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Lakshmi Durairaj, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200903757
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-07

CONDITIONS: Chronic Sinusitis
Keywords: Xylitol vs. Saline; nasal washes; sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Xylitol; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xylitol (Experimental): isotonic xylitol for sinus rinse
  Interventions: Drug: Xylitol
- Saline (Active Comparator): saline for sinus rinse
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Xylitol — 5% solution for sinus rinse
  Arms: Xylitol
Drug: Saline — saline for sinus rinse
  Other Names: Salt solution
  Arms: Saline

SUMMARY:
Is a xylitol nasal rinse better or worse than saline on patient satisfaction.

DETAILED DESCRIPTION:
In this pilot study, the investigators plan to compare the efficacy of twice daily xylitol nasal rinse with saline rinse which is the current standard, on outcomes such as quality of life and exacerbations.

ELIGIBILITY:
We now have two arms to this study.

Group I: Immunocompetent subjects with chronic rhinosinusitis

Inclusion Criteria:

* 56 Adult subjects (18 or older) presenting to the ENT(ears, nose, throat) clinics who meet the diagnosis of chronic rhinosinusitis (CRS). Definition of CRS: Presence of at least 2 of the following 4 signs/symptoms for 12 weeks or longer despite medical management:

  * Anterior and/or posterior mucopurulent drainage
  * Nasal obstruction
  * Facial pain, pressure, and/or fullness
  * Decreased sense of smell
* In addition, objective evidence of sinus mucosal disease must be demonstrated on sinus CT imaging or direct endoscopic examination.

Exclusion Criteria:

* Cystic fibrosis
* Fungal sinusitis
* Immunocompromised status (use of long term oral steroids (> 30 days), AIDS, active malignancy or chemotherapy)
* Known Ciliary disorders
* Sinonasal tumors
* Pregnancy

Group 2: CRS with antibody deficiency

* 56 Adult subjects (18 or older) presenting to the Allergy clinic who meet the diagnosis of chronic rhinosinusitis (CRS). Definition of CRS: Presence of at least 2 of the following 4 signs/symptoms for 12 weeks or longer despite medical management:

  * Anterior and/or posterior mucopurulent drainage
  * Nasal obstruction
  * Facial pain, pressure, and/or fullness
  * Decreased sense of smell
* In addition, objective evidence of sinus mucosal disease must be demonstrated on sinus CT imaging or direct endoscopic examination.

Exclusion criteria:

Cystic Fibrosis Sinonasal tumors Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Durairaj, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xylitol | Saline
Started | 27 | 26
Completed | 21 | 22
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xylitol | Saline | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (14) | 55 (17) | 54 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: SNOT-20 Scores at 12 Weeks
Description: Sinonasal outcome test is a 20 item quality of life questionnaire: Min-Max score range 0-100 The SNOT score for each patient was defined as the mean value of the response to the 20 items. The questionnaire is divided into 4 subsets, symptoms related to nose, symptoms of ear and face, sleep quality and psychological issues.
  Symptoms arereported on 100 mm visual analog scales (VASs) where 0 mm represents no symptoms and 100 mm represent "as troublesome as possible". The symptom severity is considered mild between 0 and 30, moderate from 30 to 70 and severe from 70- 100.
Time Frame: 12 weeks
Population: We initially enrolled 53 subjects but we had 10 subjects drop out of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Xylitol | Saline
Number analyzed (Participants) | 21 | 22
units on a scale | 7 (15) | 11 (16)

2. Secondary Outcome: Mean Number of Antibiotic Courses During the Study Period
Description: Mean Number of antibiotic courses for infection during the study period
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mean number of antibiotic courses during
Arm/Group | Xylitol | Saline
Number analyzed (Participants) | 21 | 22
mean number of antibiotic courses during | 1.90 (0.30) | 1.77 (0.43)

ADVERSE EVENTS:
Arm/Group | Xylitol | Saline
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes